CLINICAL TRIAL: NCT02434692
Title: A Prospective, Open-label, Multicenter Clinical Investigation to Assess the Safety and Performance of the ARGOS-IO System in Patients With Primary Open Angle Glaucoma (POAG)
Brief Title: Safety and Performance Study of the ARGOS-IO (Intraocular) System in Patients With Primary Open Angle Glaucoma (POAG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implandata Ophthalmic Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARGOS-02; CIV-13-11-011719 (Other: EUDAMED)
Record Dates: First submitted 2014-09-02; First posted 2015-05-05 (Estimated); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Primary Open Angle Glaucoma (POAG)
Keywords: Primary Open Angle Glaucoma; POAG; Glaucoma; Cataract; Surgery; Ocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm intervention ARGOS-IO system (Experimental): The ARGOS-IO Pressure sensor will be additionally implanted during local routine working procedures for cataract surgery in Patients with Primary Open Angle Glaucoma (POAG) and indicated cataract surgery.
  Interventions: Device: ARGOS-IO system

INTERVENTIONS:
Device: ARGOS-IO system — Implantation of ARGOS-IO pressure sensor after IOL placement within the cataract surgical procedure on day 0 (V01)

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the ARGOS-IO system in patients with POAG and indicated cataract surgery.

DETAILED DESCRIPTION:
This prospective, open-label, multi center, single-arm clinical investigation will enroll 22 consecutive patients.

Enrollment will be temporarily halted in case a serious adverse device effect (SADE) occurs, and Data and Safety Monitoring Board (DSMB) meeting will be conducted as soon as possible. The DSMB will then recommend whether to further continue the study as planned, or whether enrollment shall be stopped. In order to provide a complete overview of the study to the DSMB, an interim analysis will be performed after half of the study population (11-14 subjects) is enrolled with a minimum follow-up of 1 month. A conclusion for safety will be made if in total no more than 2 of the total of 22 patients experience a SADE.

The primary aim of this study is to show "safety", which will be evaluated based on the percentage of subjects who experience a SADE (="non-safety"), as defined in the primary endpoints.

The study will be declared a success if the final non-safety event rate is less than 6% (type II error rate of 0.20). The calculation is based on a design optimizing the minimum expected sample size with parameters alpha=0.05, beta=0.20, p0=0.75, p1=0.94.

ELIGIBILITY:
Inclusion Criteria:

1. Mentally competent and willing to provide written informed consent
2. Male or female aged ≥40 and ≤85 years. Female subjects of childbearing potential must be willing to use adequate contraception and must have a negative pregnancy test.
3. Diagnosis of primary open-angle glaucoma (POAG) including high pressure glaucoma (HPG), normal pressure glaucoma (NPG) and ocular hypertension (OH), as defined by the European Glaucoma Society guideline (Heijl, Treverso, et al., 2008)
4. Sufficiently controlled intraocular pressure (IOP)
5. Study eye needs to be phakic
6. Only one eye per patient may be implanted with the ARGOS-IO implant
7. Cataract surgery indicated. The medical indication for a cataract operation must be given irrespective of the study participation. Potential study patients will be solicited for participation in the clinical trial only after the patient has given consent to the cataract operation.
8. Pre-operative anterior chamber depth (ACD) ≥2.0 mm as measured from the corneal endothelium
9. Axis length >22 mm
10. Endothelial cell density of the cornea ≥2000 cells/mm²
11. Subjects able and willing to attend all scheduled visits and comply with all study procedures

Exclusion Criteria:

1. Any other type of glaucoma other than primary open-angle glaucoma as defined by inclusion criterion 3
2. Severe POAG patients with a macular degeneration and visual field loss of -20 decibels (dB) or worse in both eyes. In case of a diverse developed visual field loss, the sensor can be implanted in the worse eye for protection the better eye.
3. Exudative age-related macular degeneration, instable macular degeneration 30 days prior to inclusion, or macular edema
4. Retinal detachment
5. Corneal diseases, especially diseases affecting the corneal endothelium, e.g. Fuchs' Dystrophia
6. Diabetes mellitus
7. Existence of Marfan-Syndrome, Ehlers-Danlos-Syndrome or Weill-Marchesani-Syndrome
8. History or evidence of severe inflammatory eye diseases (i.e. uveitis, retinitis, scleritis) in one or both eyes within 6 months prior to ARGOS-IO implantation
9. Intraocular surgical procedure(s) within 6 months prior to ARGOS-IO implantation or any surgical procedure such as refractive eye surgery in the study eye that can affect the assessment of IOP by Goldmann applanation tonometry
10. History of eye tumor
11. Ocular disease other than glaucoma that may affect assessment of visual acuity and/or IOP by Goldmann applanation tonometry (choroidal hemorrhage or detachment, lens subluxation, thyroid ophthalmopathy)
12. Anterior chamber configuration that puts the subject at high risk to develop an angle closure glaucoma
13. History of extensive keloid formation
14. Severe dry eye syndrome
15. Subjects who will need to undergo ancillary procedures in the study eye at the time of implantation or during the post-operative study period
16. Any known intolerance or hypersensitivity to topical anesthetics, mydriatics, plaster or silicone (component of the device)
17. Existence of other active medical eye implant and/or other active medical implants in the head/neck region
18. Any contraindication for intraocular lens (IOL) implantation such as choroidal hemorrhage, concomitant severe eye disease, excessive vitreous loss, extremely shallow anterior chamber, microphthalmos, non-age-related cataract, posterior capsular rupture, severe corneal dystrophy, untraceable IOP, zonular separation, color vision deficiencies
19. Severe generalized disease resulting in a life expectancy shorter than a year
20. Any clinical evidence that the investigator feels would place the subject at increased risk with the placement of the device
21. Currently pregnant or breastfeeding
22. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device
23. Patients who are not suitable for the study based on the surgeon's evaluation
24. Patients unable or unwilling to understand or comply with required study procedures
25. Patients with psychiatric disorders influencing their judgement or autonomy
26. Subject and/or an immediate family member is an employee of the investigational site directly affiliated with this study, the sponsor or the contract research organization.
27. Enrollment of the fellow eye in this clinical study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Thieme, Prof., Principal Investigator — University Eye Clinic Magdeburg, Germany
Locations (11):
- Germany (11):
  - Augenklinik Universitätsklinikum Aachen, Aachen
  - Augen-Zentrum-Nordwest, Ahaus
  - Universitäts-Augenklinik Bochum, Bochum
  - Internationale Innovative Ophthalmochirurgie Breyer-Kaymak-Klabe, Düsseldorf
  - Augenklinik der SLK-Kliniken, Heilbronn
  - nordBLICK Augenklinik Bellevue, Kiel
  - Universitätsaugenklinik Magdeburg, Magdeburg
  - Augenärztliches Augenchirurgisches Zentrum (AAZ), Nuremberg
  - Klinik und Poliklinik für Augenheilkunde der Universität Rostock, Rostock
  - Knappschaftsklinikum Saar - Augenklinik, Sulzbach
  - Universitäts-Augenklinik, Tübingen

REFERENCES:
- [Derived] Mansouri K, Gillmann K, Rao HL, Weinreb RN; ARGOS-2 Study Group. Weekly and seasonal changes of intraocular pressure measured with an implanted intraocular telemetry sensor. Br J Ophthalmol. 2021 Mar;105(3):387-391. doi: 10.1136/bjophthalmol-2020-315970. Epub 2020 Jun 4. PMID 32499329
- See also: Telemetric Measurement of Intraocular Pressure via an Implantable Pressure Sensor-12-Month Results from the ARGOS-02 Trial — https://doi.org/10.1016/j.ajo.2019.09.011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from July 2014 to March 2016 in medical clinics.
Groups:
- Single-arm Intervention ARGOS-IO System: The ARGOS-IO Pressure sensor will be additionally implanted during local routine working procedures for cataract surgery in Patients with Primary Open Angle Glaucoma (POAG) and indicated cataract surgery.
  ARGOS-IO system: Implantation of ARGOS-IO pressure sensor after cataract surgery on Day 0 (V01)
Period: Overall Study
Arm/Group | Single-arm Intervention ARGOS-IO System
Started (24 patients with primary open angle glaucoma were initially enrolled. One patient was included due to a misunderstanding of the inclusion and exclusion criteria, which was noticed before the procedure. Of the 23 patients (= "Safety Set"-Group = Safety Set (SS), as specified by the protocol), 22 patients successfully received the ARGOS-IO implant (= "Single-arm intervention ARGOS-IO system"-Group = Per-Protocol-Set (PPS), as specified by the protocol) and were subjected to the follow-up visits.) | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Set: In this multicenter, open-label, single-arm, interventional clinical trial a total of 24 patients with primary open angle glaucoma were initially enrolled, 22 of whom successfully received the ARGOS-IO implant. Of the two patients, initially enrolled but not implanted with the ARGOS-IO implant, one patient was included due to a misunderstanding of the inclusion and exclusion criteria, which was noticed before the procedure. 23 patients were thus included in the safety evaluation set ("Safety Set"-Group). Due to surgical complications during cataract surgery, an implantation of the ARGOS-IO pressure sensor was not attempted in the second patient.
  Goldmann applanation tonometry (GAT) measures were compared with the sensors' IOP measures and comprehensive ophthalmic examinations at all post-operative visits (V02-V11) through 12 months.
Arm/Group | Safety Set
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 23
Number of patients who successfully received the ARGOS-IO implant [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Patients Experiencing a Device Related SAE (SADE) and Complications During Implantation
Description: Number of patients experiencing a device related SAE (SADE) and complications during the implantation of the ARGOS-IO device.
Time Frame: Day 0 to Day 360 (V01 [Implantation] to V11)
Measure: Number; unit: participants
Groups:
- Safety Set: In this multicenter, open-label, single-arm, interventional clinical trial a total of 24 patients with primary open angle glaucoma were initially enrolled, 22 of whom successfully received the ARGOS-IO implant. Of the two patients, initially enrolled but not implanted with the ARGOS-IO implant, one patient was included due to a misunderstanding of the inclusion and exclusion criteria, which was noticed before the procedure. 23 patients were thus included in the safety evaluation set ("Safety Set"-Group). Due to surgical complications during cataract surgery, an implantation of the ARGOS-IO pressure sensor was not attempted in the second patient.
Arm/Group | Safety Set
Number analyzed (Participants) | 23
participants
  SADEs | 0
  SAEs | 9
  Surgical complications | 7

2. Primary Outcome: Performance: Intraclass Correlation Between Intraocular Pressure (IOP) Measurements by GAT and the ARGOS-IO System
Description: Intraclass correlation between intraocular pressure (IOP) measurements made by GAT and the ARGOS-IO system (IOP in mmHg; starting at visit V05 as specified by the protocol) following the ICC(3,k) concordance analysis method [Choritz et al., 2019 (Telemetric Measurement of … ARGOS-02 Trial) in the "References"-section].
Time Frame: Day 30 to Day 360 (V05 to V11)
Population: All available GAT and ARGOS-IO measurements.
Measure: Number (95% Confidence Interval); unit: Intraclass correlation coefficient
Units Other Than Participants: comparisons
Groups:
- Single-arm Intervention ARGOS-IO System: In this multicenter, open-label, single-arm, interventional clinical trial, 22 patients received ARGOS-IO implants ("Single-arm Intervention ARGOS-IO System"-Group). During the 12 months following surgery, the patients returned for 10 follow-up visits consisting of comprehensive ophthalmic examinations as well as IOP measurements with the ARGOS-IO system and Goldmann Applanation Tonometry (GAT).
Arm/Group | Single-arm Intervention ARGOS-IO System
Number analyzed (Participants) | 22
Number analyzed (comparisons) | 435
Intraclass correlation coefficient | 0.789 [0.743 to 0.8717]

3. Secondary Outcome: Safety: Incidence, Nature, Severity & Seriousness of Observed AEs/ADEs.
Description: Safety evaluation based on the incidence, nature, severity and seriousness of observed adverse events and adverse device events.
Time Frame: Day 0 to Day 360 (V01 [Implantation] to V11)
Population: 168 AEs were reported, 74 AEs in 18 patients (p) were related to the ARGOS-IO device, 90 AEs in 21 p had a relationship to the medical procedure & 52 AEs in 17 p were related to other. Most common but as well expected AEs even after a standard cataract surgery were increased IOP (2 x in 14 p), anterior chamber inflammation (11x in 9 p) & anterior chamber fibrin (5 p). Pigment dispersion was described in 8 p.
Measure: Number; unit: A(D)Es
Arm/Group | Safety Set
Number analyzed (Participants) | 23
A(D)Es
  Overall number of AEs/ADEs | 168
  AEs related to medical device | 74
  AEs related to medical procedure | 90
  AEs related to other | 52

ADVERSE EVENTS:
Time Frame: Evaluation over 12 months follow-up period.
Description: SAE Definition
  That meets any of the following criteria of a serious adverse event:
  * Resulted in death, permanent damage or disability or a congenital anomaly
  * Was life threatening
  * Required hospitalization
Arm/Group | Safety Set
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=23)
Abnormal visual field test (Eye disorders) | 1 (1)
Anterior chamber fibrin (Eye disorders) | 2 (2)
Intraocular pressure increased (Eye disorders) | 2 (2)
Amaurosis fugax (Eye disorders) | 1 (1)
Corneal decompensation (Eye disorders) | 1 (1)
Cataract operation in fellow eye (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Arthritis (Immune system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=23)
Intraocular pressure increased (Eye disorders) | 12 (20)
Anterior chamber inflammation (Eye disorders) | 9 (11)
Pigment dispersion (Eye disorders) | 8 (8)
Anterior chamber fibrin (Eye disorders) | 3 (3)
Corneal endothelial cell loss (Eye disorders) | 5 (5)
Visual acuity reduced (Eye disorders) | 5 (5)
Blepharitis (Eye disorders) | 4 (4)
Corneal pigmentation (Eye disorders) | 4 (5)
Dry eye (Eye disorders) | 4 (4)
Iris prolapse (Eye disorders) | 4 (4)
Iris transillumination defect (Eye disorders) | 4 (4)
Corneal edema (Eye disorders) | 3 (3)
Macular edema (Eye disorders) | 3 (3)
Posterior capsule opafication (Eye disorders) | 3 (3)
Visual field test abnormal (Eye disorders) | 2 (2)
Conjunctival edema (Eye disorders) | 2 (2)
Corneal erosion (Eye disorders) | 2 (2)
Eye Pain (Eye disorders) | 2 (2)
Foreign body sensation in eye (Eye disorders) | 2 (2)
Glare (Eye disorders) | 2 (2)
Pupils unequal (Eye disorders) | 2 (2)
Vitreous floaters (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-02-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT02434692/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT02434692/SAP_001.pdf